CLINICAL TRIAL: NCT04232423
Title: Efficacy and Dosage of Olanzapine for Chemotherapy-induced Nausea and Vomiting Prophylaxis in Women With Gynecologic Cancers Receiving Carboplatin-based Regimen : a Double-blind, Placebo-controlled, Randomized Crossover Trial
Brief Title: Olanzapine for Chemotherapy-induced Nausea and Vomiting Prophylaxis
Acronym: OLN-EME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 162/2562
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-07

CONDITIONS: Complete Response Rate to Chemotherapy-induced Nausea and Vomiting Prophylaxis
Keywords: Olanzapine; Chemotherapy-induced nausea and vomiting; Carboplatin; Gynecologic cancer
MeSH Terms: conditions — Vomiting | interventions — Olanzapine; Tablets

STUDY DESIGN:
Intervention Model Description: A Double-Blind, Placebo-Controlled, Randomized Crossover Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- OLN 0-5-10 (Experimental): Placebo tablet in chemotherapy cycle 1, olanzapine 5 mg tablet in chemotherapy cycle 2, and olanzapine 10 mg tablet in chemotherapy cycle 3
  Interventions: Drug: Olanzapine 10 Mg ORAL TABLET; Drug: Olanzapine 5 Mg ORAL TABLET; Drug: Placebo ORAL TABLET
- OLN 5-10-0 (Experimental): Olanzapine 5 mg tablet in chemotherapy cycle 1, olanzapine 10 mg tablet in chemotherapy cycle 2, and placebo tablet in chemotherapy cycle 3
  Interventions: Drug: Olanzapine 10 Mg ORAL TABLET; Drug: Olanzapine 5 Mg ORAL TABLET; Drug: Placebo ORAL TABLET
- OLN 10-0-5 (Experimental): Olanzapine10 tablet in chemotherapy cycle 1, placebo tablet in chemotherapy cycle 2, and olanzapine 5 mg tablet in chemotherapy cycle 3
  Interventions: Drug: Olanzapine 10 Mg ORAL TABLET; Drug: Olanzapine 5 Mg ORAL TABLET; Drug: Placebo ORAL TABLET

INTERVENTIONS:
Drug: Olanzapine 10 Mg ORAL TABLET — * Olanzapine 10 mg orally, ondansetron 8 mg intravenously, and dexamethazone 8 mg intravenously 30 minutes before chemotherapeutic administration (day 1)
  * Olanzapine 10 mg orally daily and dexamethazone 8 mg orally daily on day 2, 3, 4
Drug: Olanzapine 5 Mg ORAL TABLET — * Olanzapine 5 mg orally, ondansetron 8 mg intravenously, and dexamethazone 8 mg intravenously 30 minutes before chemotherapeutic administration (day 1)
  * Olanzapine 5 mg orally daily and dexamethazone 8 mg orally daily on day 2, 3, 4
Drug: Placebo ORAL TABLET — * Placebo 1 tab orally, ondansetron 8 mg intravenously, and dexamethazone 8 mg intravenously 30 minutes before chemotherapeutic administration (day 1)
  * Placebo 1 tab orally daily and dexamethazone 8 mg orally daily on day 2, 3, 4

SUMMARY:
To investigate that olanzapine can reduced side effect about nausea and vomiting in women with gynecologic cancers receiving carboplatin-based regimen by using olanzapine and placebo

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, randomized crossover trial

ELIGIBILITY:
Inclusion Criteria:

* Women with gynecological cancer receiving carboplatin-based chemotherapeutic regimen
* ECOG performance status 0-1
* Normal bone marrow, liver, and renal functions
* Can speak and write in Thai language

Exclusion Criteria:

* Women with nausea or vomiting prior to chemotherapeutic administration
* Pregnant women
* Women with active infection
* Women with bowel obstruction
* Women with symptomatic brain metastases
* Women who received dopamine receptor antagonists within 1 week before chemotherapeutic administration
* Women who received corticosteroid within 1 week before chemotherapeutic administration
* Women with past history of chemotherapy or radiotherapy
* Women with psychiatric disorders
* Women with poor controlled diabetes mellitus
* Women who received anticonvulsant medication
* Women with history of neuroleptic malignant syndrome
* Women with history of olanzapine allergy
* Women with history of lactose intolerance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Complete response rate of chemotherapy-induced nausea and vomiting prophylaxis | 5 days after chemotherapeutic administration
  No breakthrough vomiting and no using rescue therapy

SECONDARY OUTCOMES:
Episodes of vomiting | 5 days after chemotherapeutic administration
Severity of nausea | 5 days after chemotherapeutic administration
Use of rescue drug | 5 days after chemotherapeutic administration
  using of rescue anti-emetic medication
Quality of life associated with nausea and vomiting measured using Functional Living Index-Emesis (FILE) | 5 days after chemotherapeutic administration

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand